CLINICAL TRIAL: NCT04373733
Title: A Randomised Controlled Trial of Early Intervention in Patients HospItalised With COVID-19: Favipiravir and StaNdard Care vErsEs Standard CaRe
Brief Title: Early Intervention in COVID-19: Favipiravir Verses Standard Care
Acronym: PIONEER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: NEAT ID Foundation (Other); FUJIFILM Toyama Chemical Co., Ltd. (Industry); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW002; 2020-001449-38 (EudraCT Number)
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; Coronavirus
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: Open-label parallel group randomised control trial. One trial treatment arm and one standard of care comparator arm.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir & Standard of Care (Experimental): Favipiravir: Day 1 1800mg twice per day, Days 2-10 800mg twice per day
  Interventions: Drug: Favipiravir; Other: Standard of care management
- Standard of care (Other): No trial intervention
  Interventions: Other: Standard of care management

INTERVENTIONS:
Drug: Favipiravir — Anti-viral
  Other Names: Avigan
  Arms: Favipiravir & Standard of Care
Other: Standard of care management — Standard of care management for COVID-19

SUMMARY:
Currently we do not know how best to treat patients infected with COVID-19. This study is looking at whether randomising participants to either favipiravir or to usual care, can help patients with suspected or proven COVID-19 infection.

DETAILED DESCRIPTION:
A prospective, randomised, open label study of the combined use of favipiravir and standard clinical care verses standard clinical care alone.

A computer-based software will randomise participants 1:1 to either receive favipiravir and standard medical care or standard medical care alone. The allocated medical regime will commence for 10 days.

Research blood, sputum nose swab and urine samples will be collected at baseline, as well as between day 5 and 10, and between day 14 and 28 to enable comparative analyses.

A COVID-19 antibody test will also be performed 14-28 days after randomisation. In the event of clinically indicated bronchoscopy taking place within 28 days of consent then additional bronchoscopy washing and brushing samples and paired blood sample will be taken for research purposes If a participant is discharged before one of the latter time points, they will be required to return to hospital (provided they are well enough) for the collection of repeat samples.

Participants will be closely monitored whilst taking the study medications. Participants will study exit at subject death or 28 days post-randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants: Signed informed consent
2. New admission to hospital for period expected to last ≥ 1 night
3. Suspected or confirmed COVID-19 infection

   Patients are suspected of COVID-19 infection if they have the following:

   · Influenza like illness (fever ≥37.8°C and at least one of the following respiratory symptoms, which must be of acute onset: persistent cough, hoarseness, nasal discharge or congestion, shortness of breath, sore throat, wheezing or sneezing).

   And

   · Finding from either a chest x-ray or CT suggestive of Covid-19 infection

   And

   · Alternative causes are considered unlikely
4. For women to be eligible to enter and participate in the study they should be: of non-child-bearing

   * potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   * or of child-bearing potential have a negative pregnancy test at screening and agrees to remain sexually abstinent or use a method of contraception with a failure rate of < 1% per year as indicated in Appendix B during the treatment and for a period of 7 days after the last dose. Hormonal contraceptive methods must be supplemented by a barrier method.
5. Men who are sexually active must use an adequate method of contraception as listed in Appendix B, for a period of at least 7 days after the last dose

Exclusion Criteria:

1. Pregnant or breast feeding, due to potential teratogenicity
2. Hepatic impairment - (AST or ALT > 3.5 x upper limit of normal)
3. Presently enrolled in an interventional drug study
4. Unable to take medication via the oral or nasogastric route
5. Known sensitivity Favipiravir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to a sustained clinical improvement (maintained for 24 hours) by two points on a seven-category ordinal scale or to discharge, whichever occurs first | Up to 28 days from randomisation
  Time from randomisation to a sustained clinical improvement (maintained for 24 hours) by two points on a seven-category ordinal scale or to discharge, whichever occurs first
  The seven-category ordinal scale is :
  1. Not hospitalised with resumption of normal activities
  2. Not hospitalised, but unable to resume normal
  3. Hospitalised, not requiring supplemental oxygen
  4. Hospitalised, requiring supplemental oxygen
  5. Hospitalised, requiring nasal high-flow oxygen therapy, non-invasive mechanical ventilation or both
  6. Hospitalised, requiring ECMO (Extra-corporal membrane oxygenation), invasive mechanical ventilation or both
  7. Death

SECONDARY OUTCOMES:
Clinical status on a seven-category ordinal scale (Day 7) | Day 7 from randomisation
  Clinical status of patients at given on the seven-category ordinal scale (see primary endpoint for scale)
Clinical status on a seven-category ordinal scale (Day 14) | Day 14 from randomisation
  Clinical status of patients at given on the seven-category ordinal scale (see primary endpoint for scale)
Overall survival | 28 days from randomisation
  Survival of patients to end of study
Time to improvement by two points on the NEWS score | Up to 28 days from randomisation
  Time from randomisation to improvement by two points on the NEWS score of patient condition, if maintained for 24 hours. For details of NEWS score see https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
Time to improvement by two points on the NEWS element score for temperature | Up to 28 days from randomisation
  Time from randomisation to improvement by two points on the NEWS element score for temperature, if maintained for 24 hours. For details of NEWS score see https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
Time to improvement by two points on the NEWS element score for heartrate | Up to 28 days from randomisation
  Time from randomisation to improvement by two points on the NEWS element score for heartrate, if maintained for 24 hours. For details of NEWS score see https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
Time to improvement by two points on the NEWS element score for respiratory rate | Up to 28 days from randomisation
  Time from randomisation to improvement by two points on the NEWS element score for respiratory rate, if maintained for 24 hours. For details of NEWS score see https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
Time to improvement by two points on the NEWS element score for oxygen saturation. | Up to 28 days from randomisation
  Time from randomisation to improvement by two points on the NEWS element score for oxygen saturation, if maintained for 24 hours. For details of NEWS score see https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
Admission to intensive care | Up to 28 days from randomisation
  Frequency of admission of patients to intensive care
Requirement for mechanical ventilation | Up to 28 days from randomisation
  Frequency of requirement to administer mechanical ventilation to patients
Requirement for non-invasive ventilation, continuous positive airways pressure or high-flow oxygen | Up to 28 days from randomisation
  Frequency of requirement to administer non-invasive ventilation, continuous positive airways pressure or high-flow oxygen to patients
Incidence of bacterial or fungal infection | Up to 28 days from randomisation
  Frequency of culture-confirmed bacterial or fungal infection in patients
Incidence of adverse events not directly caused by COVID-19 infection. | Up to 28 days from randomisation.
  Frequency and severity of adverse events in patients not directly attributed by clinicians to COVID-19 infection.

OTHER OUTCOMES:
Readmission to inpatient care | Up to 28 days from randomisation
  Frequency of readmission to inpatient care of patients discharged from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (6):
- Brazil (2):
  - Grupo Hospitalar Conceição, Porto Alegre
  - Fundação Oswaldo Cruz - Instituto Nacional de Infectologia Evandro Chagas (Fiocruz/INI), Rio de Janeiro
- Instituto Nacional de Ciencias Medicas y Nutricion, Salvador Zubiran, Mexico City, Mexico
- United Kingdom (3):
  - Hull University Teaching Hospitals NHS Trust - Castle Hill Hospital, Hull
  - Chelsea and Westminster Hospital, London
  - West Middlesex University Hospital, London

IPD SHARING:
Plan to Share IPD: No
Research team wishes to enable any meta-analyses of COVID-19 trials making appropriate requests. No plan to share IPD has been made at this time.

REFERENCES:
- [Derived] Shah PL, Orton CM, Grinsztejn B, Donaldson GC, Crabtree Ramirez B, Tonkin J, Santos BR, Cardoso SW, Ritchie AI, Conway F, Riberio MPD, Wiseman DJ, Tana A, Vijayakumar B, Caneja C, Leaper C, Mann B, Samson A, Bhavsar PK, Boffito M, Johnson MR, Pozniak A, Pelly M; PIONEER trial group. Favipiravir in patients hospitalised with COVID-19 (PIONEER trial): a multicentre, open-label, phase 3, randomised controlled trial of early intervention versus standard care. Lancet Respir Med. 2023 May;11(5):415-424. doi: 10.1016/S2213-2600(22)00412-X. Epub 2022 Dec 14. PMID 36528039